



# Protocol of a Thesis for partial fulfillment of M.D. degree of Orthopedic Surgery

# Title of the protocol: Total Knee Arthroplasty in conjunction with intra-operative Genicular Nerve Radio-Frequency Ablation, A randomized controlled clinical trial

Post graduate student: Assem Mohamed Mahmoud Ahmed

**Degree**: Master degree of orthopedic surgery

**Director: Professor Amr Khairy Mahmoud** 

Academic position: Professor

**Department:** Orthopedic surgery

Co-director: Professor Ibrahim Mostafa El Ganzoury

Academic position: Professor

**Department:** Orthopedic surgery

Co-director: Professor Haytham Abdelazim Mohamed

**Academic position:** Professor **Department:** Orthopedic surgery

Co-director: Dr. Ahmed Mohamed Mohasseb

**Academic position**: Assistant professor

**Department:** Orthopedic surgery

12-1-2022





## What is already known about this subject? What does this study add?

Total knee arthroplasty (TKA) is considered the gold standard management for advanced knee osteoarthritis, however around 20% of the patients still complain of persistent knee pain after the operation<sup>1</sup>. This study will add a new concept of combining genicular nerve radiofrequency ablation (GNRFA) with TKA In a hypothesis to improve functional outcome, post-operative pain and quality of life.

## 1.Introduction/Review

Total knee arthroplasty is a very common operation, and its incidence is believed to increase furthermore in the near future<sup>2</sup>. Thats why there are a lot of studies focused on improving the patient's satisfaction rate, while the unsatisfied patients remain to vary from 10%-30% without any noticeable complications<sup>3</sup>. Early post operative rehabilitation and fast track protocols showed improvement in functional outcome and pain relief but are still hindered by the patients compliance<sup>4</sup>. The idea of implementing genicular nerve radio-frequency ablation in combination with TKA rose when GNRFA showed significant improvement in patients with chronic knee osteoarthritis, studies showed pain relief up to 67% at the first 3 months, yet alone it has a very slim indications as it addresses only the biological aspect of the knee osteoarthritis without resolving the mechanical problem that will continue to progress over time<sup>5</sup>. Other studies showed positive outcome of GNRFA in cases of chronic knee pain after TKA<sup>6</sup>, <sup>7</sup>.

Given that data, combining GNRFA with TKA might give the patient a better chance to proceed with early rehabilitation programs improving the functional outcome, while decreasing postoperative pain is also considered an important factor of patients' satisfaction and quality of life enhancement.





## 2.Aim/Objectives

To compare between conventional Total Knee Arthroplasty (TKA) and Total Knee Arthroplasty (TKA) combined with intra-operative Genicular Nerve Radio-Frequency Ablation (GNRFA), concerning post-operative functional outcome and pain scores in patients with advanced knee osteoarthritis.

## 3. Methodology

- Type of the study: Randomized controlled clinical trial
- Study setting: Ain Shams University hospitals
- Study period: 24 months
- Study population: Patients with advanced knee osteoarthritis

#### Inclusion criteria:

- Both sexes
- o Age from 50-80 years old

#### **Exclusion criteria:**

- o Patients unfit for surgery
- Patients underwent previous GNRFA
- Sampling method: Convenient sample
- Sample size: 70 knees will be randomly divided by a computer-generated sequence in to 2 groups:
  - o Group A (≈35 knees): will undergo TKA
  - o Group B (≈35 knees): will undergo TKA combined with GNRFA
- Ethical considerations: will be followed by obtaining the hospital research/ethics committee approval and written informed consents from the patients.





#### • Study tools:

#### Preoperative diagnosis and evaluation:

#### Clinical Evaluation:

- History
- General examination
- Local examination (pre-operative)

#### > Radiological Evaluation:

- Plain X-ray antero-posterior standing view of the diseased knee.
- Plain X-ray lateral view of the diseased knee.

#### > Laboratory investigations:

Routine preoperative lab investigations

## Operative technique:

Patients will be operated using standard mid-vastus approach, conventional GNRFA

### Post-operative management:

- Proper antibiotic and standardized analgesics protocol will be given post-operative
- Prophylaxis against DVT
- Post-operative x-rays will be done, Plain X-ray anteroposterior and lateral view of the operated knee.





#### Follow up strategy:

Patients will be reviewed after 2 weeks to check their wounds and for sutures removal, then the follow up will be every month in the first 6 months then every 3 months till the end of the study (2 years). The follow up will include:

#### Clinical and functional assessment:

- Oxford knee score to assess the function.
- Visual analogue scale (VAS) to assess pain.
- Emotional acceptance/ Patient satisfaction.

#### > Radiological assessment:

Plain X-ray as described before at every follow up visit.

- Statistical Analysis: Statistical package for social science (SPSS 15.0.1 for windows; SPSS Inc., Chicago, IL, 2001). Data will be presented as Mean and Standard deviation (+/-SD) for quantitative parametric data, and Median and Interquartile range for quantitative non-parametric data. Frequency and percentage will be used for presenting qualitative data. Suitable analysis will be done according to the type of data obtained. P<0.05 will be considered significant.</li>
- **Statistical package:** data entry and statistical analysis of the collected data will be performed using a reliable software program.





### 4.References

- 1. Malik AT, Khan S, Ali A, Mufarrih SH, Noordin S. Total knee arthroplasty: does day of surgery matter? *Clinical Medicine Insights: Arthritis and Musculoskeletal Disorders*. 2018;11:1179544117754067.
- 2. Inacio MCS, Paxton EW, Graves SE, Namba RS, Nemes S. Projected increase in total knee arthroplasty in the United States—an alternative projection model. *Osteoarthritis and cartilage*. 2017;25(11):1797-1803.
- 3. Kim SJ, Bamne A, Song YD, Kang YG, Kim TK. Patients still wish for key improvements after total knee arthroplasty. *Knee surgery & related research*. 2015;27(1):24.
- 4. Vavro M, Ziakova E, Gazdikova K, Farkasova D. Does standard post-operative rehabilitation have its place after total knee replacement? Bratislavske lekarske listy. 2016;117(10):605-608.
- 5. Ferdinand Iannaccone D, Samuel Dixon R, Andrew Kaufman M. A review of long-term pain relief after genicular nerve radiofrequency ablation in chronic knee osteoarthritis. *Pain physician*. 2017;20:E437-E444.
- 6. Leong JF, Rani RA, bin Anuar MS, Ariff MAM, Hamdan N, Yahaya M. An Alternative Way to Relieve Neuropathic Pain After Total Knee Replacement by Genicular Nerve Radio-Frequency Ablation.
- 7. Protzman NM, Gyi J, Malhotra AD, Kooch JE. Examining the feasibility of radiofrequency treatment for chronic knee pain after total knee arthroplasty. *PM&R*. 2014;6(4):373-376.